CLINICAL TRIAL: NCT04053686
Title: A-REST (Activity to Reduce Excessive Sitting Time): a Cluster Randomised Controlled Feasibility Trial to Reduce Prolonged Sitting in Police Staff
Brief Title: An Intervention to Reduce Prolonged Sitting in Police Staff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bedfordshire (Other)
Responsible Party: Principal Investigator, Marsha Brierley, PhD Student, University of Bedfordshire
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019ISPAR008
Record Dates: First submitted 2019-07-29; First posted 2019-08-12 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Sedentary Behavior; Metabolic Syndrome; Affect; Stress, Physiological; Stress, Psychological; Musculoskeletal Pain
MeSH Terms: conditions — Sedentary Behavior; Metabolic Syndrome; Stress, Psychological; Musculoskeletal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The intervention group will aim to regularly break up participants' prolonged sitting time with three-minute incidental movement breaks every half hour at work. Support for behaviour change will include a lecture/workshop, electronic prompts, break logging, team competition, health champions, and email support.
  Interventions: Behavioral: Breaks

INTERVENTIONS:
Behavioral: Breaks — 3-min breaks every half hour at work

SUMMARY:
The primary aim of this study is to assess the feasibility of an intervention to reduce and break up prolonged sitting time in full-time police staff. The secondary aims of this study are to assess preliminary effects on patterns of sedentary behaviour (number of breaks, number of prolonged sitting bouts, average duration of prolonged sitting bouts, and total prolonged sitting duration), additional measures of sedentary behaviour (total sitting time, standing, and stepping), cardiometabolic risk markers, physiological stress (cortisol levels), physical health (self-report and postural stability), psychological wellbeing and mood, work stress (self-reported), and work performance (job satisfaction and productivity).

DETAILED DESCRIPTION:
Prolonged sedentary behaviour is associated with a higher incidence of cardiovascular disease and type 2 diabetes. A large proportion of daily sedentary time (sitting) occurs in the workplace. On average, full time office workers spend upwards of 70% of their working day seated with the majority of this time accumulated in sitting bouts ≥ 20 minutes. A recent cross-sectional investigation into the occupational characteristics of over 5,000 British police force employees reported at least 30% identifying as having mainly office-based duties. When trying to reduce prolonged sitting in the workplace, one of the most effective strategies is the use of multi-component interventions. At the present time, sedentary workplace intervention studies in the police are limited.

The primary aim of this study is to assess the feasibility of an intervention to reduce and break up prolonged sitting time at work in full-time police staff. The secondary aims of this study are to assess preliminary effects on sedentary behaviour, cardiometabolic risk markers, physiological stress, physical health, psychological wellbeing and mood, work stress, and work performance.

This has a single-arm, pre-post study design. Participants will receive a multi-component intervention to break up and reduce prolonged sitting including: a presentation/workshop, electronic support, minor environmental modifications, organisational support, and team competition. Assessments will take place at baseline and post-intervention (week 10).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 0.6 Full Time Equivalent (FTE) work hours
* Ambulatory
* Predominantly desk-based (spend on average ≥ 5-h/day seated at work by self-report)
* Own a smartphone, with ability to keep phone with them during work hours

Exclusion Criteria:

* Planned absence of two weeks or more during the intervention period
* Work part time (< 0.6 FTE)
* Health contraindications to standing and walking
* Planned relocation to another site, office or workplace
* Have personal access to an active workstation (sit-stand desk, seat cycle, treadmill desk or similar)
* Participating simultaneously in another workplace intervention (for sedentary behaviour, physical activity, diet, lifestyle, or combination thereof)
* Health contraindications to postural stability testing (e.g., injury to the lower extremities in the past six months, dizziness, or epilepsy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Feasibility - Adherence: Drop-out rates in control and intervention group | From recruitment (typically 4 weeks prior to baseline) up to study completion (typically 12 weeks)
  Analyses of drop-out rates (%) in control and intervention group.
Feasibility - Acceptability: Perceptions of the intervention | At week 11
  Asking participants' to qualitatively reflect on the intervention via semi-structured interview.

SECONDARY OUTCOMES:
Change in the number of breaks (sit-stand transitions) from sedentary time per hour (workplace and daily) | This measure will be assessed at baseline and 10 weeks. At each time point the accelerometer will be worn for 7 days.
  Participants will wear a thigh-based accelerometer/inclinometer (ActivPAL3), which provides a well established measure of sit-stand transitions.
Change in sitting time accrued in prolonged bouts (≥ 30 minutes) (workplace and daily) | This measure will be assessed at baseline and 10 weeks. At each time point the accelerometer will be worn for 7 days.
  Participants will wear a thigh-based accelerometer/inclinometer (ActivPAL3), which provides a well established measure of sitting time accrued in prolonged bouts (≥ 30 minutes).
Change in the average duration (minutes) of prolonged sitting bouts (≥ 30 minutes) (workplace and daily) | This measure will be assessed at baseline and 10 weeks. At each time point the accelerometer will be worn for 7 days.
  Participants will wear a thigh-based accelerometer/inclinometer (ActivPAL3), which provides a well established measure of the average duration (minutes) of prolonged sitting bouts (≥ 30 minutes).
Change in the number of prolonged sitting bouts (≥ 30 minutes) (workplace and daily) | This measure will be assessed at baseline and 10 weeks. At each time point the accelerometer will be worn for 7 days.
  Participants will wear a thigh-based accelerometer/inclinometer (ActivPAL3), which provides a well established measure of the number of prolonged sitting bouts (≥ 30 minutes).
Change in the total duration (minutes) of sitting time (workplace and daily) | This measure will be assessed at baseline and 10 weeks. At each time point the accelerometer will be worn for 7 days.
  Participants will wear a thigh-based accelerometer/inclinometer (ActivPAL3), which provides a well established measure of sitting time.
Change in step count (workplace and daily) | This measure will be assessed at baseline and 10 weeks. At each time point the accelerometer will be worn for 7 days.
  Participants will wear a thigh-based accelerometer/inclinometer (ActivPAL3), which provides a well established measure of step count.
Change in total stepping time (in minutes) (workplace and daily) | This measure will be assessed at baseline and 10 weeks. At each time point the accelerometer will be worn for 7 days.
  Participants will wear a thigh-based accelerometer/inclinometer (ActivPAL3), which provides a well established measure of total stepping time (in minutes).
Change in total standing time (in minutes) (workplace and daily) | This measure will be assessed at baseline and 10 weeks. At each time point the accelerometer will be worn for 7 days.
  Participants will wear a thigh-based accelerometer/inclinometer (ActivPAL3), which provides a well established measure of total standing time (in minutes).
Weight (kg) | Baseline and at week 11
  Changes in weight via Tanita scale.
Body mass index (BMI) | Baseline and at week 11
  Changes in BMI will be computed by dividing participants' weight (in kilograms) by their height (in metres) squared.
Waist circumference (cm) | Baseline and at week 11
  Changes in waist circumference will be assessed by tape measure.
Body fat % | Baseline and at week 11
  Changes in body fat percentage will be assessed via a bioelectric impedance spectroscopy device.
Body fat mass (kg) | Baseline and at week 11
  Changes in body fat mass via a bioelectric impedance spectroscopy device.
Lean body mass (kg) | Baseline and at week 11
  Changes in lean body mass via a bioelectric impedance spectroscopy device.
Blood pressure (mmHg) | Baseline and at week 11
  Changes in blood pressure measured via electronic sphygmomanometer.
Fasted blood cholesterol (mg/dL) | Baseline and at week 11
  Changes in total, high density lipoprotein (HDL), and low density lipoprotein (LDL) cholesterol measured via fasting blood tests using a Cholestech machine.
Fasted blood triglycerides (mg/dL) | Baseline and at week 11
  Changes in triglycerides measured via fasting blood tests using a Cholestech machine.
Fasted blood glucose (mg/dL) | Baseline and at week 11
  Changes in glucose levels measured via fasting blood tests using a Cholestech machine.
Salivary cortisol (nmol/L) | Baseline and at week 11. At each time point saliva samples will be collected at 7 time points over the course of one day.
  Changes in the cortisol awakening response and diurnal cortisol levels will be assessed via saliva samples (provided by chewing on a cotton swab for 60secs) collected seven times over the course of one day.
Nordic musculoskeletal questionnaire | Baseline and at week 11
  The Nordic musculoskeletal questionnaire is comprised of 40 forced-choice questions pertaining to low back, neck, shoulder and general physical complaints most often experienced in the work setting. A visual diagram aids the viewer by labelling the nine regions of the body referred to in the questionnaire. Acceptable reliability for this tool has been demonstrated.
Postural sway velocity (mm/s) | Baseline and at week 11
  Change in postural sway velocity (bipedal-eyes-open, bipedal-eyes-closed, unipedal-eyes-open, unipedal-eyes-closed) will be evaluated via dynamic plantar pressure sensor (RS Footscan).
Postural sway range (mm) | Baseline and at week 11
  Change in postural sway range (bipedal-eyes-open, bipedal-eyes-closed, unipedal-eyes-open, unipedal-eyes-closed) will be evaluated via dynamic plantar pressure sensor (RS Footscan).
International Physical Activity Questionnaire short form (IPAQ) | Baseline and at week 11
  Changes in self-reported physical activity and total sitting time. The International Physical Activity Questionnaire short form (IPAQ) measures self-reported physical activity and sitting time in the last seven days. Participants are asked to report frequency of participation (0-7 days) and duration of activity on one of those days (in hours and minutes). The IPAQ has demonstrated acceptable reliability and validity in measuring activity in the last seven days.
Marshall sitting questionnaire | Baseline and at week 11
  The Marshall sitting questionnaire has five questions that measure self-reported domain-specific sitting time (hours and minutes) on weekend days and weekdays. This questionnaire has good reliability and validity for sitting time on weekdays and weekend days.
Warwick-Edinburgh mental well-being scale (WEMWBS) | Baseline and at week 11
  The Warwick-Edinburgh mental well-being scale (WEMWBS) is a 14-item questionnaire used to assess various aspects of positive mental health (e.g., "I've been feeling optimistic about the future"). Participants are asked to rate their experience of each wellbeing statement between 1 and 5 (1 = none of the time and 5 = all of the time). Item scores are then combined to provide a total score (between 14 - 70). The higher the score the better the overall mental wellbeing. For intervention purposes, a change in the total score of 3-8 points between two time points may be considered a "meaningful change".
Positive and negative affect schedule (PANAS) | Baseline and at week 11
  Changes in self-reported mood via the positive and negative affect schedule (PANAS) consisting of two 10-item subscales to measure positive and negative affect (i.e., mood). A number of words that describe different feelings and emotions (e.g., "interested", "distressed", "excited") are presented and participants are asked to indicate on a 5-point scale to what extent over the past week they have felt these feelings/emotions (1 = very slightly or not at all and 5 = extremely). These scales are internally consistent with very good convergent and discriminant correlations.
  Negative Affect subscale Item scores on the negative affect scale are then combined to provide a total score (between 10 - 50). The higher the score the more negative emotions experienced.
  Positive Affect subscale Item scores on the positive affect scale are then combined to provide a total score (between 10 - 50). The higher the score the more positive emotions experienced.
Operational police stress questionnaire (PSQ-Op) | Baseline and at week 11
  Changes in ratings of 20 operational stressors for police (PSQ-Org). Participants will be asked to rate items on "how much stress it has caused you over the past 6 months" using a 7-point Likert scale (1 = no stress at all and 7 = a lot of stress). Item scores are then combined to provide a total score (between 20 - 140). The higher the score the worse the stress level. This instrument has demonstrated acceptable reliability and validity for measuring police-specific occupational stressors.
Organisational police stress questionnaire (PSQ-Org) | Baseline and at week 11
  Changes in ratings of 20 organisational stressors for police (PSQ-Org). Participants will be asked to rate items on "how much stress it has caused you over the past 6 months" using a 7-point Likert scale (1 = no stress at all and 7 = a lot of stress). Item scores are then combined to provide a total score (between 20 - 140). The higher the score the worse the stress level. This instrument has demonstrated acceptable reliability and validity for measuring police-specific occupational stressors.
Job satisfaction | Baseline and at week 11
  Changes in self-reported job satisfaction and will be evaluated via a single-item questionnaire ("How satisfied are you with your job in general?") assessed on a 7-point Likert scale (1 = dissatisfied and 7 = extremely satisfied). A higher score represents more satisfaction with one's job.
Job performance | Baseline and at week 11
  Changes in self-reported job performance will be evaluated via a single-item questionnaire ("How well do you think you have performed in your job recently?") with a 7-point Likert scale (1 = very poorly and 7 = extremely well). A higher score represents a more positive assessment of job performance.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bailey, PhD, Principal Investigator — University of Bedfordshire
Locations (1):
- University of Bedfordfordshire, Bedford, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided